CLINICAL TRIAL: NCT04061837
Title: To Evaluate the Effectiveness and Safety of MitralStitch Mitral Valve Repair System - a Clinical Application of New Technology
Brief Title: MitralStitch Mitral Valve Repair System for Mitral Regurgitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Jian Yang, Deputy chief surgeon, Xijing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJ-20190823
Record Dates: First submitted 2019-08-14; First posted 2019-08-20 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MitralStitch repair system (Experimental): Experimental group is allocated to use novel mitral valve repair system manufactured by Hangzhou Valgen Medtech Co., Ltd
  Interventions: Device: MitralStitch

INTERVENTIONS:
Device: MitralStitch — With transesophageal echocardiographic guidance,implanting ePTFE sutures as artificial chordae or ege-to-ege repair using MitralStitch Mitral Valve Repair System

SUMMARY:
The main objective is to assess the effectiveness and safety of the MitralStitch repair system in patients with moderate to severe and severe mitral regurgitation.

ELIGIBILITY:
Inclusion Criteria:

1. The age of patient is ≥18yrs;
2. Severe mitral regurgitation patients (The area of central regurgitation exceeds 40% of left atrial area or holosystolic eccentric regurgitation; VC≥0.07cm；regurgitant volume ≥60ml；RF ≥50%; EROA≥0.4cm2 (Satisfy any condition).
3. LVESD≤60mm, LVEF≥25%, small incision surgery of chest can be tolerated.
4. The subject was informed of the clinical application nature of the new technology and agreed to participate in all requirements of the clinical application of the new technology, signed the ICF and agreed to complete the follow-up and the inspection required during the follow-up period.

Exclusion Criteria:

1. Subject who are pregnant, lactating or scheduled to pregnant during the period of the clinical new technology.
2. Subjects with active endocarditis or rheumatic mitral valve disease.
3. Life expectancy <1 year for cardiac or other malignant tumors.
4. Participate in other clinical trial
5. In the judgment of the investigator, subjects had poor acceptance of chemotherapy, and they cannot complete the trial as required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence rate of major adverse event after 30 days of the intervention | 30days
  The occurrence of complications associated with any device or operation, including but not limited to: death, emergency surgery, severe pericardial tamponade requiring pericardiac puncture or surgery, bleeding, and surgically related stroke.

SECONDARY OUTCOMES:
The success of device | Immediately after repair
  The MitralStitch mitral valve repair system reaches the mitral valve and implant the chord and withdraw the system successfully.
The success rate of operation | Before discharge, an average of 7 days
  Mitral regurgitation was less than moderate before discharge.
Incidence of major adverse events after device implantation | 12months
  There were no major adverse events associated with device or operation within 12 months of device implantation.
The classification of mitral regurgitation | 1/6/12 months
  Mild: No mitral regurgitation or the centricity regurgitation area is smaller than the 20% of left atrial area.
  Moderate: The area of centricity regurgitation is upper than 40%, lower than 60% of the left atrial area; VC≥0.7cm; regurgitant volume≥60ml； RF≥50%; EROA≥0.4cm².
  Severe: The area of centricity regurgitation is upper than 40% of the left atrial area or systolic eccentric regurgitation.

CONTACTS AND LOCATIONS:
Overall Officials: Shiqiang Yu, Principal Investigator — Xijing Hospital; Jian Yang, Study Director — Xijing Hospital
Locations (1):
- Department of Cardiovascular Surgery of Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No